CLINICAL TRIAL: NCT04045054
Title: Home-based Team Transitional Telecare to Optimize Mobility and Physical Activity in Recently Hospitalized Older Veterans
Brief Title: Home-based Transitional Telecare for Older Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Ann Arbor Healthcare System (U.S. Federal Agency)
Collaborators: University of Michigan (Other); Michigan Health Endowment Fund (Other)
Responsible Party: Principal Investigator, Neil Alexander, Director, Ann Arbor Geriatric Research Education and Clinical Center, VA Ann Arbor Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AWD004365
Record Dates: First submitted 2019-05-17; First posted 2019-08-05 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Telemedicine; Veterans Health; Physical Activity; Mobility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): The Link Team follows up with the participants for 6 months after they discharge from the hospital
  Interventions: Behavioral: Link Team

INTERVENTIONS:
Behavioral: Link Team — A VA home care Link Team (clinical pharmacist, social worker, physical activity trainer) provides the intervention based on a conceptual model of home care as a bridge between hospital and home, in which three interconnected domains determine short-term and long-term outcomes: medical complexity (e.g., medication management), social complexity (e.g., caregiving, environment), and functional impairment (e.g., mobility, physical activity). The Link Team provides support and assessment for each domain, and will use tablet technology and wearable sensors in the home to gather patient data and facilitate communication. At the end of formal home care services, the Link Team provides patient-centered care in: 1) support for the the Veteran and caregiver in the event of changes in medical condition or medications and social or caregiver stressors; and 2) coaching to the Veteran and the caregiver during this transition period to optimize functional mobility and physical activity.

SUMMARY:
The project focuses on supporting home care in the post-hospitalization period (Home Health Phase), and then further optimizing the older Veterans' recovery of mobility and physical activity in the transition back to the home/community (Follow-up Phase).

DETAILED DESCRIPTION:
Medicare-funded home care bridges gaps in the transition of patients from hospital to home; yet, it is a bridge with gaps of its own, having limited communication with both the discharging hospital physician and the receiving primary care provider and having limited knowledge of the longitudinal medical history of the patient. Once home care is completed, there is often no plan of continued support to transition the older Veteran back to optimal home/community function.

In the Home Health Phase, a VA-home care Link Team (physician, clinical pharmacist, social worker, and physical activity trainer) will provide immediate communication/coordination between the VA Ann Arbor Healthcare System (VAAAHS) and home care agencies contracted by VAAAHS. The intervention is based on a conceptual model of home care as a bridge between hospital and home, in which three interconnected domains determine short-term and long-term outcomes: medical complexity (e.g., medication management), social complexity (e.g., caregiving, environment), and functional impairment (e.g., mobility, physical activity). The VA Link Team will provide support and assessment for each domain. The team will use telemedicine technology and wearable sensors in the home to gather patient data and facilitate communication between the patient, health care providers, and the Link Team. The Follow-up Phase begins at the end of formal home care services, when the Link Team will provide patient-centered care in two ways: 1) support for the the Veteran and caregiver in the event of changes in medical condition or medications as well as social or caregiver stressors; and 2) coaching to the Veteran and the caregiver during this transition period to optimize functional mobility and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Under VA Ann Arbor Healthcare System (VAAAHS) primary care practitioner (PCP) oversight.
* Recently discharged from inpatient hospitalization.
* Received inpatient (pre-discharge) physical therapy evaluation and have identified rehabilitation goals for care to be provided in the home.
* Identified caregiver who agrees to participate and who will be the key link if the Veteran is unable to care for himself or has memory problems.

Exclusion Criteria:

* Require highly specialized equipment or therapy (e.g. rehabilitation for spinal cord injury, prosthesis training following leg amputation).
* Have active mental health conditions (e.g. paranoia) that may interfere with program participation.
* Require strict bed rest (e.g. long-term extensive wound healing needs) or strict use of a wheelchair.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Telemedicine Encounters | 1 year
  Number of successful telemedicine encounters is measured for each participant.
Successful Telemedicine Encounter Rate | 1 year
  Percentage of successful telemedicine encounters is measured for each participant.

SECONDARY OUTCOMES:
Remote Short Portable Performance Battery (rSPPB) | (1) Baseline; (2) Up to 6 months; (3) Up to 1 year.
  The rSPPB, based on the widely used SPPB measures of walking speed, multiple chair stands, and standing balance, will be performed with caregiver standby assist while the Veteran is viewed via the tablet camera.
Wearable sensors | (1) Baseline; (2) Up to 6 months; (3) Up to 1 year.
  Physical activity will be measured over a seven day period with a research grade sensor, the activPAL3VT.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Alexander, MD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alexander NB, Phillips K, Wagner-Felkey J, Chan CL, Hogikyan R, Sciaky A, Cigolle C. Team VA Video Connect (VVC) to optimize mobility and physical activity in post-hospital discharge older veterans: baseline assessment. BMC Geriatr. 2021 Sep 22;21(1):502. doi: 10.1186/s12877-021-02454-w. PMID 34551725